CLINICAL TRIAL: NCT03524664
Title: Parent Emotion Socialization and Child Emotion Regulation in FASD
Brief Title: A Study of Parent and Child Emotions in Fetal Alcohol Spectrum Disorder (FASD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Christie Petrenko, Research Associate, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RSRB69545; R34AA025717 (NIH)
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Results first posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Fetal Alcohol Spectrum Disorders
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed "tuning in to kids" intervention (No Intervention): Children with fetal alcohol spectrum disorder and their parents
- "Tuning in to kids" intervention (Experimental): Children with fetal alcohol spectrum disorder and their parents
  Interventions: Behavioral: Tuning In to kids intervention

INTERVENTIONS:
Behavioral: Tuning In to kids intervention — The Tuning Into Kids Program involves:
  * Meeting in a small group with other caregivers raising children with FASD.
  * 8-week program that meets weekly for 2 hours at Mt. Hope Family Center or other community location.
  * Learn and practice an approach of responding to children's emotions and behavior.
  Arms: "Tuning in to kids" intervention

SUMMARY:
The purpose of this study is to learn about the emotion regulation skills of children with fetal alcohol spectrum disorders (FASD) and different strategies that may improve these skills. This study is also testing whether a training program taught to caregivers is helpful.

Children will be asked to:

* Complete a brief measure of verbal and nonverbal problem-solving skills.
* Play two computer games.
* Have their heart rate measured while completing a task that is designed to be mildly disappointing. Two ECG pads are placed on the chest with a small recorder.
* Play or relax with study staff while you are finishing caregiver activities.

Caregivers will be asked to complete interviews and questionnaires about:

* the child's background, including any past stressful experiences
* the child's behavior and how s/he handles emotions
* caregiver views on the child's emotions and their own
* caregiver relationship with the child
* Stress caregivers experience as a parent

DETAILED DESCRIPTION:
Children with fetal alcohol spectrum disorders (FASD) have high rates of mental health problems and incur physical and mental health expenditures that are 9 times higher than other children. These mental health problems contribute to poor social adjustment for children with FASD and result in considerable emotional and financial burden for families. Emotion regulation is a core area of impairment in FASD and is implicated in most mental health disorders. Research on empirically validated interventions for children with FASD is limited. Results from two interventions targeting emotion regulation in FASD demonstrate that child-focused interventions are insufficient to habilitate children's emotion regulation to adaptive levels. Research is needed to identify alternate targets for intervention (e.g., parent training, environmental modifications) to improve the emotion regulation difficulties of children with FASD.

This study investigates a novel intervention target to improve the emotion regulation and adaptive functioning of children with FASD. Research with other populations provides ample evidence for the impact of parent emotion socialization on the development of child emotion regulation and other outcomes. In addition, studies demonstrate that parent emotion socialization is amendable to intervention and results in improved child and parent outcomes. However, no studies have investigated the emotion socialization practices utilized by parents of children with FASD or whether interventions targeting parent emotion socialization result in improved child emotion regulation and behavior in this population.

This study will address this critical gap by initiating an empirical test of a promising emotion-focused intervention, Tuning In To Kids (TIK), with families raising children with FASD. Results from this initial efficacy trial will determine whether parent emotion socialization is a promising intervention target for this population. Consistent with a developmental psychopathology perspective, multi-level data from the efficacy trial will be leveraged to test theorized associations between parent emotion socialization and child emotion regulation and identify possible factors contributing to individual differences. These results will inform possible intervention adaptations for this population and provide the necessary foundation for larger-scale efficacy trials. The long-term goals of this research are to better understand the complex factors influencing emotion regulation in children with FASD and improve mental health interventions and outcomes for this population.

ELIGIBILITY:
Inclusion Criteria:

Families will be eligible for the study if they:

* Have a child between the age of 4 and 12 with a formal diagnosis of an FASD based on the Revised 2016 Hoyme criteria (Hoyme et al., 2016)
* The child is in some form of out of home care (e.g., adoptive, foster, relative, or other legal guardian)
* The child has resided with the primary caregiver for at least a year and be expected to remain in that placement for at least 6 months (study duration).

Exclusion Criteria:

* A history of other genetic, neurological, or significant medical conditions, traumatic brain injury, serious psychiatric illness or disability that would preclude data collection
* Child has a moderate to severe intellectual disability (IQ < 55)
* Child or caregiver has insufficient proficiency in English
* Caregiver is a biological parent of the child with FASD

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mt. Hope Family Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petrenko CLM, Kautz-Turnbull C, Rockhold MN, Handley ED, Havighurst SS, Toth SL. Results of a pilot randomized controlled trial of Tuning in to Kids for children with FASD in nonbiological parent care. Alcohol Clin Exp Res (Hoboken). 2025 Oct;49(10):2349-2364. doi: 10.1111/acer.70153. Epub 2025 Aug 29. PMID 40884006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Families were primarily recruited from a University Medical Center Diagnostic Clinic for fetal alcohol spectrum disorders. Providers gave potentially eligible families a flyer about the study. Families then contacted the study team to complete screening over the phone.
Pre-assignment Details: 118 families were screened for eligibility. A total of 2 has incomplete screening, 10 were excluded for not meeting inclusion criteria, 4 declined to participate, 13 were not able to schedule baseline assessments, and 2 withdrew or were lost to contact after baseline assessments, but before randomization. A total of 87 families were randomized to study arm.
Groups:
- Delayed "Tuning in to Kids" Intervention: Children with fetal alcohol spectrum disorder and their parents
  Received the Tuning in to Kids intervention about 5-6 months after randomization.
- "Tuning in to Kids" Intervention: Children with fetal alcohol spectrum disorder and their parents
  Tuning In to kids intervention: The Tuning Into Kids Program involves:
  * Meeting in a small group with other caregivers raising children with FASD.
  * 8-week program that meets weekly for 2 hours at Mt. Hope Family Center or other community location, or virtually (during COVID-19 pandemic).
  * Learn and practice an approach of responding to children's emotions and behavior.
Period: Overall Study
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Started | 33 | 54
Completed Allocated Condition | 33 | 37 (Completing 5 or more of the 8 sessions was defined as completion of the intervention program. A total of 7 participants started but discontinued intervention program. Ten did not start the program)
Immediate Post-Intervention Follow-up Assessments (T2) | 32 | 45
3-month Post-Intervention Follow-up Assessments (T3) | 28 | 39
Completed | 28 | 39 (Completing 5 or more of the 8 sessions was defined as completion of the program)
Not Completed | 5 | 15
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 4 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention | Total
Number analyzed (Participants) | 33 | 54 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] — Parent age
  years | 48.16 (9.93) | 46.72 (9.97) | 47.28 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants] — Caregiver Sex
  Participants
    Female | 32 | 53 | 85
    Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Caregiver Ethnicity
  Participants
    Hispanic or Latino | 2 | 1 | 3
    Not Hispanic or Latino | 29 | 47 | 76
    Unknown or Not Reported | 2 | 6 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants] — Caregiver Race
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 3 | 7 | 10
    White | 28 | 42 | 70
    More than one race | 1 | 0 | 1
    Unknown or Not Reported | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 33 | 54 | 87
Child Age [Mean (Standard Deviation); unit: years] | 8.18 (2.89) | 7.54 (2.52) | 7.78 (2.67)
Child Sex at Birth [Count of Participants; unit: Participants]
  Female | 11 | 20 | 31
  Male | 22 | 34 | 56
Child Race [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 14 | 19
  White | 22 | 26 | 48
  More than One Race | 2 | 8 | 10
  Unknown or Not Reported | 3 | 5 | 8
Child Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 24 | 41 | 65
  Unknown or Not Reported | 5 | 9 | 14

OUTCOME MEASURES:

1. Primary Outcome: Parent Awareness of Own Emotion Score for Sadness at Baseline and Immediate Post-intervention (8 Weeks)
Description: The meta emotion interview is a semi-structured interview administered to parents about their own experience of anger and sadness and their feelings, attitudes, and behaviors toward their children's anger and sadness. Interviews can be analyzed quantitatively using a checklist rating system. The Revised Meta-Emotion coding system uses a 5-point Likert scale (1= strongly disagree to 5= strongly agree) with which coders rate each item based on both the content and the way parents talk about emotions. The parent awareness sub-scale for sadness includes 9 items; sub-scale score is a sum of items with a total range of 9 to 45. A higher score reflects greater parental awareness of their sadness.
Time Frame: baseline to immediate post-intervention (8 weeks)
Population: Outcome data analyzed for those with complete data at both timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 30 | 43
score on a scale
  Baseline (T1) | 32.73 (0.84) | 32.37 (0.70)
  Immediate Post-Intervention (T2) | 32.20 (0.67) | 32.47 (0.56)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Repeated measures ANOVA; Test type: Superiority; p = .523, ANOVA — The threshold for statistical significance was p = 0.05; F(1,71) = 0.411, p =.523

2. Primary Outcome: Parent Acceptance of Own Expression Score for Sadness at Baseline and Immediate Post-intervention (8 Weeks)
Description: The meta emotion interview is a semi-structured interview administered to parents about their own experience of anger and sadness and their feelings, attitudes, and behaviors toward their children's anger and sadness. Interviews can be analyzed quantitatively using a checklist rating system. The Revised Meta-Emotion coding system uses a 5-point Likert scale (1= strongly disagree to 5= strongly agree) with which coders rate each item based on both the content and the way parents talk about emotions. The parent acceptance of expressivity sub-scale for sadness includes 8 items; sub-scale score is a sum of items with a total range of 8 to 40. A higher score reflects greater acceptance of emotion expression for sadness.
Time Frame: baseline to immediate post-intervention (8 weeks)
Population: Outcome data analyzed for those with complete data at both timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 30 | 43
score on a scale
  Baseline (T1) | 26.07 (0.59) | 25.35 (0.49)
  Immediate Post-intervention (T2) | 26.83 (0.65) | 25.05 (0.55)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Repeated measures ANOVA; Test type: Superiority; p = .173, ANOVA — The threshold for statistical significance was p = 0.05; F(1,71)=1.89, p=.173

3. Primary Outcome: Parent Regulation of Own Emotions Score for Sadness at Baseline and Immediate Post-intervention (8 Weeks)
Description: The meta emotion interview is a semi-structured interview administered to parents about their own experience of anger and sadness and their feelings, attitudes, and behaviors toward their children's anger and sadness. Interviews can be analyzed quantitatively using a checklist rating system. The Revised Meta-Emotion coding system uses a 5-point Likert scale (1= strongly disagree to 5= strongly agree) with which coders rate each item based on both the content and the way parents talk about emotions. The parent sub-scale for regulation of their own sadness includes 6 items; sub-scale score is a sum of items with a total range of 6 to 30. A higher score reflects better parent regulation of their sadness.
Time Frame: baseline to immediate post-intervention (8 weeks)
Population: Outcome data analyzed for those with complete data at both timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 30 | 43
score on a scale
  Baseline (T1) | 23.43 (0.48) | 22.11 (0.40)
  Immediate Post-Intervention (T2) | 23.47 (0.42) | 23.14 (0.35)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Outcome data analyzed for those with complete data at both timepoints; Test type: Superiority; p = .140, ANOVA — The threshold for statistical significance was p = 0.05; F(1,71)=2.23, p=.140

4. Primary Outcome: Parent Awareness of Child Emotion Score for Sadness at Baseline and Immediate Post-intervention (8 Weeks)
Description: The meta emotion interview is a semi-structured interview administered to parents about their own experience of anger and sadness and their feelings, attitudes, and behaviors toward their children's anger and sadness. Interviews can be analyzed quantitatively using a checklist rating system. The Revised Meta-Emotion coding system uses a 5-point Likert scale (1= strongly disagree to 5= strongly agree) with which coders rate each item based on both the content and the way parents talk about emotions. The parent awareness of child's sadness sub-scale includes 8 items; sub-scale score is a sum of items with a total range of 8 to 40. A higher score reflects greater parental awareness of their child's sadness.
Time Frame: baseline to immediate post-intervention (8 weeks)
Population: Outcome data analyzed for those with complete data at both timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 30 | 42
score on a scale
  Baseline (T1) | 29.40 (0.78) | 29.48 (0.66)
  Immediate Post-Intervention (T2) | 29.97 (0.71) | 29.86 (0.60)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Outcome data analyzed for those with complete data at both timepoints; Test type: Superiority; p = 0.845, ANOVA — The threshold for statistical significance was p = 0.05; F(1,70)=.039, p=0.845

5. Primary Outcome: Parent Acceptance of Child's Emotion Score for Sadness at Baseline and Immediate Post-intervention (8 Weeks)
Description: The meta emotion interview is a semi-structured interview administered to parents about their own experience of anger and sadness and their feelings, attitudes, and behaviors toward their children's anger and sadness. Interviews can be analyzed quantitatively using a checklist rating system. The Revised Meta-Emotion coding system uses a 5-point Likert scale (1= strongly disagree to 5= strongly agree) with which coders rate each item based on both the content and the way parents talk about emotions. The parent acceptance of their child's sadness sub-scale includes 6 items; sub-scale score is a sum of items with a total range of 6 to 30. A higher score reflects greater acceptance of their child's sadness.
Time Frame: baseline to immediate post-intervention (8 weeks)
Population: Outcome data analyzed for those with complete data at both timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 30 | 42
score on a scale
  Baseline (T1) | 21.17 (0.67) | 19.98 (0.56)
  Immediate Post-Intervention (T2) | 21.33 (0.64) | 21.29 (0.54)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Outcome data analyzed for those with complete data at both timepoints; Test type: Superiority; p = .147, ANOVA — The threshold for statistical significance was p = 0.05; F(1,70)=2.147, p=.147

6. Primary Outcome: Parent Emotion Coaching Score for Sadness at Baseline and Immediate Post-intervention (8 Weeks)
Description: The meta emotion interview is a semi-structured interview administered to parents about their own experience of anger and sadness and their feelings, attitudes, and behaviors toward their children's anger and sadness. Interviews can be analyzed quantitatively using a checklist rating system. The Revised Meta-Emotion coding system uses a 5-point Likert scale (1= strongly disagree to 5= strongly agree) with which coders rate each item based on both the content and the way parents talk about emotions. The parent emotion coaching sub-scale for sadness includes 6 items; sub-scale score is a sum of items with a total range of 6 to 30. A higher score reflects greater use of emotion coaching when their child is sad.
Time Frame: baseline to immediate post-intervention (8 weeks)
Population: Outcome data analyzed for those with complete data at both timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 30 | 42
score on a scale
  Baseline (T1) | 21.33 (0.64) | 20.14 (0.54)
  Immediate Post-Intervention (T2) | 21.03 (0.61) | 20.45 (0.52)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Outcome data analyzed for those with complete data at both timepoints; Test type: Superiority; p = .429, ANOVA — The threshold for statistical significance was p = 0.05; F(1,70)=.633, p=.429

7. Primary Outcome: Child Regulation Score for Sadness at Baseline and Immediate Post-intervention (8 Weeks)
Description: The meta emotion interview is a semi-structured interview administered to parents about their own experience of anger and sadness and their feelings, attitudes, and behaviors toward their children's anger and sadness. Interviews can be analyzed quantitatively using a checklist rating system. The Revised Meta-Emotion coding system uses a 5-point Likert scale (1= strongly disagree to 5= strongly agree) with which coders rate each item based on both the content and the way parents talk about emotions. The child regulation sub-scale for sadness includes 7 items; sub-scale score is a sum of items with a total range of 7 to 35. A higher score reflects better child regulation of sadness.
Time Frame: baseline to immediate post-intervention (8 weeks)
Population: Outcome data analyzed for those with complete data at both timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 30 | 42
score on a scale
  Baseline (T1) | 23.20 (0.65) | 23.74 (0.55)
  Immediate Post-Intervention (T2) | 24.10 (0.64) | 23.43 (0.54)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Outcome data analyzed for those with complete data at both timepoints; Test type: Superiority; p = .208, ANOVA — The threshold for statistical significance was p = 0.05; F(1,70)=1.618, p=.208

8. Primary Outcome: Parent Awareness of Own Emotion Score for Anger at Baseline and Immediate Post-intervention (8 Weeks)
Description: The meta emotion interview is a semi-structured interview administered to parents about their own experience of anger and sadness and their feelings, attitudes, and behaviors toward their children's anger and sadness. Interviews can be analyzed quantitatively using a checklist rating system. The Revised Meta-Emotion coding system uses a 5-point Likert scale (1= strongly disagree to 5= strongly agree) with which coders rate each item based on both the content and the way parents talk about emotions. The parent awareness sub-scale for anger includes 9 items; sub-scale score is a sum of items with a total range of 9 to 45. A higher score reflects greater parental awareness of their own anger.
Time Frame: baseline to immediate post-intervention (8 weeks)
Population: Outcome data analyzed for those with complete data at both timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 31 | 42
score on a scale
  Baseline (T1) | 33.74 (0.65) | 33.12 (0.56)
  Immediate Post-intervention (T2) | 34.10 (0.54) | 34.31 (0.46)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Outcome data analyzed for those with complete data at both timepoints; Test type: Superiority; p = .300, ANOVA — The threshold for statistical significance was p = 0.05; F(1,71)=1.09, p=.300

9. Primary Outcome: Parent Acceptance of Own Expression Score for Anger at Baseline and Immediate Post-intervention (8 Weeks)
Description: The meta emotion interview is a semi-structured interview administered to parents about their own experience of anger and sadness and their feelings, attitudes, and behaviors toward their children's anger and sadness. Interviews can be analyzed quantitatively using a checklist rating system. The Revised Meta-Emotion coding system uses a 5-point Likert scale (1= strongly disagree to 5= strongly agree) with which coders rate each item based on both the content and the way parents talk about emotions. The parent acceptance of their anger expression sub-scale includes 8 items; sub-scale score is a sum of items with a total range of 8 to 40. A higher score reflects greater parental acceptance of their own anger expression.
Time Frame: baseline to immediate post-intervention (8 weeks)
Population: Outcome data analyzed for those with complete data at both timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 31 | 42
score on a scale
  Baseline (T1) | 24.65 (0.66) | 25.12 (0.56)
  Immediate Post-Intervention (T2) | 25.65 (0.54) | 24.69 (0.46)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Outcome data analyzed for those with complete data at both timepoints; Test type: Superiority; p = .099, ANOVA — The threshold for statistical significance was p = 0.05; F(1,71)=2.79, p=.099

10. Primary Outcome: Parent Regulation of Own Emotions Score for Anger at Baseline and Immediate Post-intervention (8 Weeks)
Description: The meta emotion interview is a semi-structured interview administered to parents about their own experience of anger and sadness and their feelings, attitudes, and behaviors toward their children's anger and sadness. Interviews can be analyzed quantitatively using a checklist rating system. The Revised Meta-Emotion coding system uses a 5-point Likert scale (1= strongly disagree to 5= strongly agree) with which coders rate each item based on both the content and the way parents talk about emotions. The parent regulation sub-scale for anger includes 6 items; sub-scale score is a sum of items with a total range of 6 to 30. A higher score reflects better parental regulation of their own anger.
Time Frame: baseline to immediate post-intervention (8 weeks)
Population: Outcome data analyzed for those with complete data at both timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 31 | 42
score on a scale
  Baseline (T1) | 21.52 (0.51) | 20.71 (0.44)
  Immediate Post-Intervention (T2) | 21.81 (0.50) | 22.24 (0.43)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Outcome data analyzed for those with complete data at both timepoints; Test type: Superiority; p = .105, ANOVA — The threshold for statistical significance was p = 0.05; F(1,71)=2.70, p=.105

11. Primary Outcome: Parent Awareness of Child Emotion Score for Anger at Baseline and Immediate Post-intervention (8 Weeks)
Description: The meta emotion interview is a semi-structured interview administered to parents about their own experience of anger and sadness and their feelings, attitudes, and behaviors toward their children's anger and sadness. Interviews can be analyzed quantitatively using a checklist rating system. The Revised Meta-Emotion coding system uses a 5-point Likert scale (1= strongly disagree to 5= strongly agree) with which coders rate each item based on both the content and the way parents talk about emotions. The parent awareness of their child's anger sub-scale includes 8 items; sub-scale score is a sum of items with a total range of 8 to 40. A higher score reflects greater awareness of their child's anger.
Time Frame: baseline to immediate post-intervention (8 weeks)
Population: Outcome data analyzed for those with complete data at both timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 31 | 42
score on a scale
  Baseline (T1) | 31.48 (0.58) | 31.17 (0.50)
  Immediate Post-Intervention (T2) | 31.10 (0.53) | 31.07 (0.46)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Repeated measures ANOVA; Test type: Superiority; p = .699, ANOVA — The threshold for statistical significance was p = 0.05; F(1,71)=0.15, p=.699

12. Primary Outcome: Parent Acceptance of Child's Emotion Score for Anger at Baseline and Immediate Post-intervention (8 Weeks)
Description: The meta emotion interview is a semi-structured interview administered to parents about their own experience of anger and sadness and their feelings, attitudes, and behaviors toward their children's anger and sadness. Interviews can be analyzed quantitatively using a checklist rating system. The Revised Meta-Emotion coding system uses a 5-point Likert scale (1= strongly disagree to 5= strongly agree) with which coders rate each item based on both the content and the way parents talk about emotions. The parent acceptance of their child's anger sub-scale includes 6 items; sub-scale score is a sum of items with a total range of 6 to 30. A higher score reflects greater parental acceptance of their child's anger.
Time Frame: baseline to immediate post-intervention (8 weeks)
Population: Outcome data analyzed for those with complete data at both timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 31 | 42
score on a scale
  Baseline (T1) | 16.71 (0.69) | 16.91 (0.59)
  Immediate Post-Intervention (T2) | 16.94 (0.66) | 17.07 (0.56)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Repeated measures ANOVA; Test type: Superiority; p = .945, ANOVA — The threshold for statistical significance was p = 0.05; F(1,71)=0.005, p=.945

13. Primary Outcome: Parent Emotion Coaching Score for Anger at Baseline and Immediate Post-intervention (8 Weeks)
Description: The meta emotion interview is a semi-structured interview administered to parents about their own experience of anger and sadness and their feelings, attitudes, and behaviors toward their children's anger and sadness. Interviews can be analyzed quantitatively using a checklist rating system. The Revised Meta-Emotion coding system uses a 5-point Likert scale (1= strongly disagree to 5= strongly agree) with which coders rate each item based on both the content and the way parents talk about emotions. The parent emotion coaching sub-scale for anger includes 6 items; sub-scale score is a sum of items with a total range of 6 to 30. A higher score reflects greater use of emotion coaching of the child's anger.
Time Frame: baseline to immediate post-intervention (8 weeks)
Population: Outcome data analyzed for those with complete data at both timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 31 | 42
score on a scale
  Baseline (T1) | 20.10 (0.66) | 19.88 (0.56)
  Immediate Post-Intervention (T2) | 20.26 (0.57) | 20.24 (0.49)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Repeated measures ANOVA; Test type: Superiority; p = .767, ANOVA — The threshold for statistical significance was p = 0.05; F(1,71)=0.088, p=.767

14. Primary Outcome: Child Regulation Score for Anger at Baseline and Immediate Post-intervention (8 Weeks)
Description: The meta emotion interview is a semi-structured interview administered to parents about their own experience of anger and sadness and their feelings, attitudes, and behaviors toward their children's anger and sadness. Interviews can be analyzed quantitatively using a checklist rating system. The Revised Meta-Emotion coding system uses a 5-point Likert scale (1= strongly disagree to 5= strongly agree) with which coders rate each item based on both the content and the way parents talk about emotions. The child regulation sub-scale for anger includes 7 items; sub-scale score is a sum of items with a total range of 7 to 35. A higher score reflects better child emotion regulation.
Time Frame: baseline to post-intervention (8 weeks)
Population: Outcome data analyzed for those with complete data at both timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 31 | 42
score on a scale
  Baseline (T1) | 18.61 (0.72) | 18.31 (0.62)
  Immediate Post-Intervention (T2) | 18.71 (0.73) | 18.05 (0.63)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Repeated measures ANOVA; Test type: Superiority; p = .682, ANOVA — The threshold for statistical significance was p = 0.05; F(1,71)=.0.17, p=.682

15. Primary Outcome: Proportion of Observed Emotion Coaching Statements Using the Family Narrative Task at Baseline and Immediate Post-intervention (8 Weeks)
Description: The Family Narrative Task is a parent-child interaction task assessing how parents communicate about emotions with their children. Parents are instructed to engage the child in a conversation about three emotional events in turn: a positive family experience, a difficult family experience, and a time when the child misbehaved. Interactions are videotaped and coded for content and function using the Family Emotion Communication Scoring System, Revised. Emotion coaching (e.g., "I could tell you were mad because you walked away," "How did you feel when that happened?") and dismissing (e.g., "It wasn't anything to get upset over," abrupt change in topic) is coded. The proportion of emotion coaching statements across all three scenarios made versus total statements is calculated. Higher scores reflect greater proportion of emotion coaching statements made.
Time Frame: baseline to immediate post-intervention (8 weeks)
Population: Outcome data analyzed for those with complete data at all timepoints. During the COVID-19 pandemic, interview measures were completed over Zoom with research staff, whereas questionnaires were sent electronically to families to complete. Completion rate of questionnaires and observational tasks was lower.
Measure: Mean (Standard Error); unit: proportion of statements
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 16 | 28
proportion of statements
  Baseline (T1) | 0.045 (0.012) | 0.052 (.009)
  Immediate Post-Intervention (T2) | 0.039 (0.011) | 0.046 (0.008)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Repeated measures ANOVA; Test type: Superiority; p = .960, ANOVA — The threshold for statistical significance was p = 0.05; F(1,42)=0.003, p=.960

16. Primary Outcome: Proportion of Observed Emotion Dismissing Statements Using the Family Narrative Task at Baseline and Immediate Post-intervention (8 Weeks)
Description: The Family Narrative Task is a parent-child interaction task assessing how parents communicate about emotions with their children. Parents are instructed to engage the child in a conversation about three emotional events in turn: a positive family experience, a difficult family experience, and a time when the child misbehaved. Interactions are videotaped and coded for content and function using the Family Emotion Communication Scoring System, Revised. Emotion coaching (e.g., "I could tell you were mad because you walked away," "How did you feel when that happened?") and dismissing (e.g., "It wasn't anything to get upset over," abrupt change in topic) is coded. The proportion of emotion dismissing statements across all three scenarios versus total statements is calculated, with higher proportions reflecting more use of emotion dismissing statements.
Time Frame: baseline to immediate post-intervention (8 weeks)
Population: Outcome data analyzed for those with complete data at all timepoints. During the COVID-19 pandemic, interview measures were completed over Zoom with research staff, whereas questionnaires were sent electronically to families to complete. Completion rate of observation tasks and questionnaires was lower.
Measure: Mean (Standard Error); unit: proportion of statements
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 16 | 28
proportion of statements
  Baseline (T1) | 0.014 (0.005) | 0.011 (0.004)
  Immediate Post-intervention (T2) | 0.006 (0.003) | 0.006 (0.002)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Repeated measures ANOVA; Test type: Superiority; p = .643, ANOVA — The threshold for statistical significance was p = 0.05; F(1,42)=0.218, p=.643

17. Primary Outcome: Child Emotion Regulation Using the Emotion Regulation Checklist at Baseline, Immediate Post-intervention, and 3-month Post-intervention Follow-up
Description: The Emotion Regulation Checklist is a 24-item parent report questionnaire assessing children's affect lability (e.g., "exhibits wide mood swings," "is easily frustrated") and emotion regulation (e.g., "is empathetic towards others," "can say when s/he is feeling sad, angry, fearful, or afraid"). This assessment is 24 items rated by the parent on a 4 point scale of never to always given at baseline, 8 and 20 weeks. There are 12 items of lability and 12 items of emotion regulation. Items are summed for each sub-scale. For the emotion regulation sub-scale the score ranges from 12-48 with higher scores reflecting better emotion regulation.
Time Frame: baseline, immediate post-intervention (8 weeks), 3-month post-intervention follow-up
Population: Outcome data analyzed for those with complete data at all timepoints. During the COVID-19 pandemic, interview measures were completed over Zoom with research staff, whereas questionnaires were sent electronically to families to complete. Completion rate of questionnaires was lower.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 21 | 26
score on a scale
  Baseline (T1) | 24.14 (0.66) | 23.36 (0.60)
  Immediate Post-Intervention (T2) | 23.22 (0.77) | 23.81 (0.69)
  Three-Months Post-Intervention (T3) | 23.43 (0.68) | 23.54 (0.61)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Repeated measures ANOVA; Test type: Superiority; p = .118, ANOVA — The threshold for statistical significance was p = 0.05; Time X Group F(2,90)=2.19, p.118

18. Primary Outcome: Child Lability/Negativity Using the Emotion Regulation Checklist at Baseline, Immediate Post-intervention, and 3-month Post-intervention Follow-up
Description: The Emotion Regulation Checklist is a 24-item parent report questionnaire assessing children's affect lability (e.g., "exhibits wide mood swings," "is easily frustrated") and emotion regulation (e.g., "is empathetic towards others," "can say when s/he is feeling sad, angry, fearful, or afraid"). This assessment is 24 items rated by the parent on a 4 point scale of never to always given at baseline, 8 and 20 weeks. There are 12 items of lability and 12 items of emotion regulation. Item scores are summed for each sub-scale. For the lability/negativity sub-scale, the score ranges from 12-48 with higher scores reflecting worse lability/negativity.
Time Frame: baseline, immediate post-intervention (8 weeks), 3-month post-intervention follow-up
Population: as for outcome 17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 21 | 26
score on a scale
  Baseline (T1) | 38.61 (1.37) | 40.64 (1.23)
  Immediate Post-Intervention (T2) | 38.89 (1.60) | 41.00 (1.44)
  Three-Month post-Intervention (T3) | 39.38 (1.77) | 40.74 (1.59)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Repeated measures ANOVA; Test type: Superiority; p = .800, ANOVA — The threshold for statistical significance was p = 0.05; Time x Group F(2,90)=.223, p=.800

19. Primary Outcome: Intensity of Disruptive Behaviors Using the Eyberg Child Behavior Inventory at Baseline, Immediate Post-intervention, and 3-month Post-intervention Follow-up
Description: The Eyberg Child Behavior Inventory is a 36-item scale assessing the intensity of disruptive behaviors in children. Parents rate each item on a 7 point scale. This is then converted into a standardized score with a "T-score" with mean of 50 and standard deviation of 10. Higher scores reflecting more problems. This is given at baseline, immediate post-intervention (8 weeks) and 3-month post-intervention follow-up. Scores are considered clinically elevated when T>60.
Time Frame: baseline, immediate post-intervention (8 weeks), 3-month post-intervention follow-up
Population: as for outcome 17
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
Number analyzed (Participants) | 20 | 28
T-score
  Baseline (T1) | 64.00 (1.61) | 66.68 (1.36)
  Immediate Post-Intervention (T2) | 63.20 (1.59) | 66.75 (1.34)
  Three-Month Post-Intervention (T3) | 63.40 (1.85) | 66.32 (1.57)
Statistical Analysis 1: Comparison: Delayed "Tuning in to Kids" Intervention vs "Tuning in to Kids" Intervention; Repeated measures ANOVA; Test type: Superiority; p = .863, ANOVA — The threshold for statistical significance was p = 0.05; Group x Time F(2,92)=0.148, p=.863

ADVERSE EVENTS:
Time Frame: Baseline, immediate post-intervention (8 weeks), and 3-month post-intervention follow-up.
Description: Adverse events in children with FASD or their caregivers could include aggression or violence towards others, maltreatment, self-harm or suicidality, or the need for inpatient hospitalization. However, these occurrences are unlikely to be a direct consequence of participation in the caregiver intervention or study. These were not systematically assessed but procedures were in place to assess risk and respond appropriately if they arose. No adverse events were detected or reported.
Arm/Group | Delayed "Tuning in to Kids" Intervention | "Tuning in to Kids" Intervention
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/54
Other Adverse Events (participants affected / at risk) | 0/33 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT03524664/Prot_SAP_000.pdf
  • Informed Consent Form: Caregiver Consent Form (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT03524664/ICF_001.pdf
  • Informed Consent Form: Permission Form (child in foster care) (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT03524664/ICF_002.pdf
  • Informed Consent Form: Child Assent (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT03524664/ICF_003.pdf